CLINICAL TRIAL: NCT06354322
Title: Physiopathological Investigation of Unclassified GENotypes of Autoinflammatory Diseases and AA Amyloidosis
Brief Title: Unclassified GENotypes of Autoinflammatory Diseases and AA Amyloidosis
Acronym: IPHYGENI MAI
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230630
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: AA Amyloidosis; Autoinflammatory Disease
Keywords: Autoinflammatory disease; AA amylosis; Functional explorations; Unclassified genotypes
MeSH Terms: conditions — AA amyloidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMC, fibroblasts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients to be studied
- Control patients

SUMMARY:
Patients with autoinflammatory diseases (AID) have recurrent episodes of systemic inflammation accompanied by nonspecific elevation of blood inflammation markers typically absent between attacks. A complication of autoinflammatory diseases is AA amyloidosis, which can lead to renal failure and dialysis. Advances in genetic analysis have led to the identification of new autoinflammatory diseases and thus new pathophysiological pathways.

However, genetic analyses are sometimes confronted with results that are difficult to interpret. These are the Variants of Unknown Significance, for which genetic analysis alone does not allow to determine if the genetic mutation is responsible for the symptoms.

genetic analysis sometimes has limitations in the diagnosis of AID which can only be overcome by pathophysiological studies of the variants found.

DETAILED DESCRIPTION:
The study aim to explore variants of undetermined significance in major and minor patients with unclassified autoinflammatory disease or AA amyloidosis of undetermined etiology by studying their pathogenicity.

National multicenter research: internal medicine department of Tenon Hospital, pediatric department of Versailles Hospital and pediatric dermatology department of Necker Enfants Malades Hospital in Paris

Samples will be collected at the inclusion visit or at subsequent visits of the patient to the department during a blood draw performed as part of routine care by a registered nurse.

The total volume of the sample will be 24 mL per 6 month period maximum, and will not exceed In case of skin involvement of the auto-inflammatory disease, a skin biopsy may be performed as part of the patient's follow-up care.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients to be studied:

* Patients over 18 years of age with the capacity to give express free and informed consent and;
* Minor patients under 18 years of age with both parents or legal guardians giving consent;
* Patients with unclassified IAD or AA amyloidosis of undetermined etiology;
* Patients followed in one of the study departments;
* Patients weighing more than 15 kg.

Inclusion criteria for control patients:

* Patients over 18 years of age with the capacity to give free and informed express consent;
* Patients with IAD classified with well-defined international criteria or ;
* Patients who have undergone cosmetic surgery or blood donors).

Exclusion Criteria:

* Patients unable to give express free and informed consent;
* Subjects under guardianship, curatorship or safeguard of justice;
* Subjects who do not speak French;
* Subjects unable to answer questions or express themselves;
* Patients weighing less than 15 kg;
* Patients without social security coverage

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Major and minor patients with unclassified autoinflammatory disease or AA amyloidosis of undetermined etiology
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2039-02 (Estimated); Study Completion 2039-02 (Estimated)

PRIMARY OUTCOMES:
Exploration of VUS in AutoInflammatory Diseases | Up to 4 years
  To explore variants of undetermined significance (VUS)in patients with unclassified autoinflammatory disease or AA amyloidosis of undetermined etiology by studying their pathogenicity.

SECONDARY OUTCOMES:
Pathophysiology of Autoinflammatory Diseases | Up to 4 years
  To improve the knowledge on the pathophysiology of Autoinflammatory Diseases: to determine the role of new inflammation pathways in AutoInflammatory Diseases
Role of other innate immune cells in AutoInflammatory Diseases | Up to 4 years
  Evaluate the role of other innate immune cells (neutrophils, mast cells...) and their mediators
Improve knowledge of AA amyloidosis | Up to 4 years
  Improve knowledge of AA amyloidosis, a complication of autoinflammatory diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Service médecine interne-Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: No